CLINICAL TRIAL: NCT05589272
Title: TDCS-potentiated Generalization of Cognitive Training in the Rehabilitation of Long COVID Symptoms
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Didn't receive IRB approval
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 30319 protocol
Record Dates: First submitted 2022-10-19; First posted 2022-10-21 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Post-acute Sequelae SARS-CoV-2 Infection (PASC)

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive training + active-tDCS (Experimental): Cognitive training + active-tDCS 4 times per week (20 minutes per session, each (~25cm²; current density = 0.08 mA/cm²); anode on left dorsolateral prefrontal cortex F3, cathode on right dorsolateral prefrontal cortex F4) for four weeks.
  Interventions: Other: Active tDCS
- Cognitive training + sham-tDCS (Sham Comparator): Cognitive training + sham-tDCS 4 times per week (20 minutes per session, each ~25cm²; current density = 0.08 mA/cm²); anode on left dorsolateral prefrontal cortex F3, cathode on right dorsolateral prefrontal cortex F4) for four weeks.
  Interventions: Other: Sham tDCS

INTERVENTIONS:
Other: Active tDCS — cognitive training + active-tDCS tDCS twice a day (two 13 minute sessions per day, each 2mA / 25cm² = 0.08 current density; anode on left dorsolateral prefrontal cortex F3, cathode on right dorsolateral prefrontal cortex F4) for five consecutive days.
  Arms: Cognitive training + active-tDCS
Other: Sham tDCS — cognitive training + sham-tDCS tDCS twice a day (two 13 minute sessions per day, each 2mA / 25cm² = 0.08 current density; anode on left dorsolateral prefrontal cortex F3, cathode on right dorsolateral prefrontal cortex F4) for five consecutive days.
  Arms: Cognitive training + sham-tDCS

SUMMARY:
The overarching goals of this study are to employ cognitive testing to understand how transcranial direct current stimulation (tDCS), when used concurrently with cognitive training tasks, can affect cognitive impairment symptoms in individuals with long COVID, or post-acute sequelae SARS-CoV-2 infection (PASC), and to examine variability in response between active and sham tDCS treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide consent and comply with study procedures
* Age 18 to 60 years old
* Estimated IQ within the specified range (70 <= IQ E <= 115)
* Current post-acute sequelae SARS-CoV-2 infection (PASC) as defined by the National Center for Health Statistics post-COVID-19 conditions survey ((Long COVID 2022), including impaired cognition symptoms, for at least 3 months post-infection
* Ability to participate in four weekly 40' training sessions over four weeks and participate in two assessments
* English speaking

Exclusion Criteria:

* Any medical condition or treatment with neurological sequelae (e.g. stroke, tumor, loss of consciousness >30 min, concussion involving hospital admission, HIV)
* Contraindications for tDCS (e.g. history of seizures)
* Five or more sessions of neuromodulation (such as tDCS) or cognitive training in the past 6 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Cognitive improvement effects of WM training with active tDCS vs. sham | baseline and post-test assessment, 4 weeks
  shown by WM task progression and performance on cognitive testing measures
Generalization of cognitive effects of active tDCS vs. sham | baseline and post-test assessment, 4 weeks
  includes effect on PASC-related cognitive impairment symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No